CLINICAL TRIAL: NCT05206825
Title: Evaluation of Electrocardiography Performed With Mobile ECG Devices in Cardiac Patients and Healthy Volunteers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Sponsor
Other Study IDs: RNN/172/20/KE
Record Dates: First submitted 2022-01-12; First posted 2022-01-25 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-01

CONDITIONS: Cardiac Arrhythmia
Keywords: Electrocardiogram; Mobile ECG
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Electrocardiography is one of most basic laboratory tests in cardiology. Novel mobile ECG are becoming popular. The investigators aim to compare typical electrocardiographic measurements obtained with mobile ECG devices (Alivecor Kardia and Alivecor Cardia 6L) and 12-leads standard ECG (gold standard). The recordings will be compared by cardiologist paying special attention to heart rhythm disturbances, components of ECG curve and quality of recording.

DETAILED DESCRIPTION:
Electrocardiography is one of most basic laboratory tests in cardiology. Novel mobile ECG are becoming popular. The investigators aim to compare typical electrocardiographic measurements obtained with mobile ECG devices (Alivecor Kardia and Alivecor Cardia 6L) and 12-leads standard ECG (gold standard). The recordings will be compared by cardiologist paying special attention to heart rhythm disturbances, components of ECG curve and quality of recording.

ECG evaluation will include: rhythm description, measurements of mean RR, PR, QRS, QT, QTc and ST-T description. Additionally inter/intraventricular conduction abnormalities are to be determined from 12-leads ECG and approximate from mobile ECG recordings.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for electrocardiography
* Informed consent to participate in the study
* The possibility of self-registration of a mobile ECG (no physical and mental restrictions)

Exclusion Criteria:

* Not willing or incapable to give written informed consent.
* Lack of willingness to cooperate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with cardiac diseases,hospitalized in Department of Electrocardiology Medical University of Lodz as well as healthy volunteers will be enrolled to the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
ECG Tracing Quality | Once: Day 0-3 after entry to the study.
  Evaluation of quality of ECG tracings obtained with different electrocardiographs
Cardiac Rhythm Determination | Once: Day 0-3 after entry to the study.
  Defining a rhythm of the patient based on recorder tracings.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Electrocardiology Medical University of Lodz, Lodz, Poland